CLINICAL TRIAL: NCT04365998
Title: Use of "BUBOLight®" Device as an Innovative Phototherapy Device for the Treatment of Newborn's Jaundice. A Monocentric, Descriptive Pilot Study, for the Feasibility, Safety and Tolerance of the BUBOLight® Device
Brief Title: BUBOLight®, a New Phototherapy Device for the Treatment of the Newborn's Jaundice
Acronym: BUBO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018_68; 2019-A01417-50 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-04-15; First posted 2020-04-28 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Neonatal Jaundice
Keywords: jaundice; phototherapy; medical device; newborn
MeSH Terms: conditions — Jaundice, Neonatal; Jaundice

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BUBOLight® Device (Experimental)
  Interventions: Device: BUBOLight® Device

INTERVENTIONS:
Device: BUBOLight® Device — 1 session of phototherapy with BUBOLight® device during 4 hours.
  Other Names: Phototherapy device with light emitting fabrics.

SUMMARY:
About 50% of full-term newborns and 80% of premature infants develop jaundice which is due to hyperbilirubinemia. In the majority of cases, jaundice disappears naturally without treatment within three weeks of birth, but the bilirubin level may remain too high, which can lead to a serious neurological disease: kernicterus. To avoid this, a therapeutic management must be instituted, and in some cases, one or more phototherapy sessions (PT) may be prescribed.

The aim of this trial is to evaluate the safety and level of satisfaction of parents and healthcare team with one innovative device for phototherapy BUBOLight® included two removable strips of luminous textile incorporating optical fibers.

10 newborns requiring phototherapy, will be illuminated during four hours in one session of PT Bilirubin levels is taken at the start of phototherapy H0 and Controls are made at H+6 hours.

ELIGIBILITY:
Inclusion Criteria:

* At time of birth, infant is > 35 weeks gestation
* Presence of jaundice confirmed by measurement of bilirubin (transcutaneous bilirubinometer)
* Total bilirubinemia rate requiring phototherapy according to National Institute for Health and Clinical Excellence.
* Weight ≥2.500kg
* Judged in good health by the investigator following the clinical examination and the medical data (absence of perinatal asphyxia, antibiotic treatment, respiratory disorders)
* Absence of fœto-maternal rhesus incompatibility or Kell

Exclusion Criteria:

* Newborn already treated with phototherapy
* Febrile state with body temperature > 37.8°C
* Total bilirubinaemia level is equal or excess 100 μmol / L of the indication of phototherapy.
* Patient whose jaundice is due to haemolysis, obstruction functional or anatomical.
* Minor relative
* Newborn requiring exchange transfusion
* Newborn with congenital erythropoietic porphyria or a family history of porphyria.
* Patient requiring treatment other than phototherapy

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2020-10-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of related adverse events (Safety) | at the begin of phototherapy (baseline, H0)
  Safety is defined as the ability to tolerate 4 hours of phototherapy without - Hyperthermia greater than or equal to 38.5 °C
  * Hypothermia less than or equal to 36 °C
  * Desaturation in O2 lower than 90% for more than 15 seconds
  * Heart rate greater than 160 / min at calm or less than 80 / min for more than 15 seconds
  * Allergic contact reaction grade ≥3
Number of related adverse events (Safety) | at 2 hours after the beginning of phototherapy (H2)
  Safety is defined as the ability to tolerate 4 hours of phototherapy without - Hyperthermia greater than or equal to 38.5 °C
  * Hypothermia less than or equal to 36 °C
  * Desaturation in O2 lower than 90% for more than 15 seconds
  * Heart rate greater than 160 / min at calm or less than 80 / min for more than 15 seconds
  * Allergic contact reaction grade ≥3
Number of related adverse events (Safety) | at the end of phototherapy exposure (H4)
  Safety is defined as the ability to tolerate 4 hours of phototherapy without - Hyperthermia greater than or equal to 38.5 °C
  * Hypothermia less than or equal to 36 °C
  * Desaturation in O2 lower than 90% for more than 15 seconds
  * Heart rate greater than 160 / min at calm or less than 80 / min for more than 15 seconds
  * Allergic contact reaction grade ≥3

SECONDARY OUTCOMES:
Blood bilirubin rate | Baseline and 2 hours after the end of phototherapy (H4+2 hours)
  Bilirubin lowering rate
Transcutaneous bilirubin rate | Baseline (H0) and 2 hours after the end of phototherapy (H4+2 hours)
  Bilirubin lowering rate
EDIN (Newborn Pain and Discomfort Scale) | Baseline (H0) and 2 hours after the end of phototherapy (H4+2 hours)
  Variation of the EDIN score between the beginning and 2 hours after phototherapy Minimum value = 0 and maximum value = 15. Above 5 pain is probable, below 5 pain is more likely to be discomfort than pain.
Perceptions of parents with the use of device | 2 hours after the end of phototherapy (H4+2 hours)
  Validated survey at the end of treatment (comfort, heat, humidity, ease of breastfeeding, proximity and possibility of contact with the baby)
Perceptions of the health team with the use of the device | 2 hours after the end of phototherapy (H4+2 hours)
  Validated survey at the end of treatment (comfort, heat, humidity, ease of breastfeeding, proximity and possibility of contact with the baby)

CONTACTS AND LOCATIONS:
Overall Officials: Thameur Rakza, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Jeanne de Flandre Chu Lille, Lille, France

REFERENCES:
- [Result] Lecomte F, Thecua E, Ziane L, Deleporte P, Duhamel A, Vamour C, Mordon S, Rakza T. Phototherapy Using a Light-Emitting Fabric (BUBOLight) Device in the Treatment of Newborn Jaundice: Protocol for an Interventional Feasibility and Safety Study. JMIR Res Protoc. 2021 May 25;10(5):e24808. doi: 10.2196/24808. PMID 34032584